CLINICAL TRIAL: NCT00821483
Title: Phase 3 Study to Assess the Efficacy and Safety of Frovatriptan
Brief Title: A Double Blind Placebo-controlled, Parallel Group Study to Assess the Efficacy and Safety of Frovatriptan in the Acute Treatment of Migraine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SK Chemicals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FRESH
Record Dates: First submitted 2009-01-12; First posted 2009-01-13 (Estimated); Last update posted 2013-04-18 (Estimated); Status verified 2013-04

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — frovatriptan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1: placebo (Placebo Comparator)
  Interventions: Drug: Frovatriptan
- 2 Frovatriptan (Active Comparator)
  Interventions: Drug: Frovatriptan

INTERVENTIONS:
Drug: Frovatriptan — 2.5mg, qd

SUMMARY:
The purpose of this study is:

1. To compare the efficacy of a single dose of Frovatriptan 2.5 mg with that of placebo in acute treatment of up to one migraine attract
2. To assess recurrence rate between two group
3. To assess the safety and tolerability

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 to 65 years
2. The patients must have a history of migraine according to the criteria of the Headache Classification Committee of the International Headache Society(IHS), over the previous 1 year. The patient must have experienced one to eight moderate or severe migraine attacks(with or without aura) each month over at least the previous two months
3. Onset of migraine disease must have occurred before the patients was 50 years of age
4. Able and willing to sign informed consent, and able and willing to comply with study procedures, including the completion of diary cards.

Exclusion Criteria:

1. Pregnant or lactating females, or women intend to become pregnant or breast feed during the study period, or women of childbearing potential not using adequate contraception. Females of reproductive potential must have a negative pregnancy test at screening
2. Clinically significant renal dysfunction(creatinine≥2.0mg/dl) or hepatic dysfunction(ALT,AST≥2 ULN)
3. Patients with clinically significant abnormal ECGs or with resting diastolic blood pressure above 95mmHg
4. Patients with clinically significant cardiovascular or cerebrovascular disease
5. Patients with a history of clinically relevant allergy, including allergy to triptan
6. Previous treatment with Frovatriptan at any time or treatment with an investigational drug within 30 days before screening visit
7. Patients with a diagnosis of vertebrobasilar or hemiplegic(prolonged atypical aura) migraine(IHS criteria)
8. Potentially unco-operative patients, those unable to provide informed consent, and those unable to complete the diary
9. patients who habitually abuse headache medication including ergotamine-containing compounds, and patients with a history of alcohol and/or medicine abuse, in the Investigator's opinion
10. Patients who are not able to tell that they are having a migraine headache
11. Patients who have 15 or more headache days per month, on average, or those taking symptomatic medication for headaches on more than two days per week, on average
12. Treatment with a monoamine-oxidase inhibitor(MAOI) within two weeks of the screening visit
13. Patients who are taking prophylactic migraine medication, unless dose has been stabilized for 30 days and it expected to continue for the duration of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2006-11; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
A comparison between Frovatriptan and placebo for the proportion of patients who have complete(grade 0) or almost complete(grade 1) relief of headache at 2 hours after taking Frovatriptan | at 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Sun U Kwon, professor, Principal Investigator — Department of Neurology, Asan Medical Center, University of Ulsan